CLINICAL TRIAL: NCT01633281
Title: A Study of Acupuncture for Bortezomib or Thalidomide -Induced Peripheral Neuropathy in Patients With Multiple Myeloma or Lymphoma
Brief Title: Acupuncture for Peripheral Neuropathy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: poor recruitment and expiry of funding
Sponsor: Singapore General Hospital (Other)
Collaborators: National Neuroscience Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Acupuncture 001
Record Dates: First submitted 2012-06-29; First posted 2012-07-04 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Peripheral Neuropathy Grade 2 or Greater
Keywords: peripheral neuropathy; acupuncture; Bortezomib; Thalidomide
MeSH Terms: conditions — Peripheral Nervous System Diseases | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- acupuncture treatment (Experimental)
  Interventions: Procedure: acupuncture

INTERVENTIONS:
Procedure: acupuncture — Ten sessions of acupuncture at 2x per week over 5 weeks will be given to patients. The acupuncture points include a standard set of obligatory points and additional points based on symptoms.

SUMMARY:
A significant proportion (up to 60%) of myeloma patients treated with Bortezomib or thalidomide or both develop significant peripheral neuropathy (PN). Standard of care for this complication include drugs like gabapentin or pregabalin, which relieve symptoms only partially. PN of grade II or above mandates reduction in dose or frequency of Bortezomib or thalidomide, which may compromise treatment outcome. This clinical study explores whether, by intervening early in its course using acupuncture, progression of PN can be reversed, stabilized or retarded thereby allowing continuation of treatment on schedule.

DETAILED DESCRIPTION:
1. The acupuncture treatment will start after patients have received at least 3 weeks of Gabapentin or Pregabalin at adequate dose without improvement in PN
2. Two sessions of acupuncture per week, each of 30minutes duration, will be administered for a total of 10 sessions over 5 weeks. The needling will be done by the designated acupuncturist for all patients, delivered with electrical stimulation at a defined frequency.
3. A fixed set of acupoints will be applied which include both local and distant points, based on both symptoms of PN and classification of TCM syndrome. Some degree of flexibility with addition or reduction of acupoints is allowed based on clinical indication. The acupoints needled each session will be recorded.
4. Assessment of efficacy 4.1 Objective response : A complete neurological examination will be done at commencement of acupuncture and at end of acupuncture.

In addition, a full nerve conduction test will be done at beginning of acupuncture and at the end of 10 sessions of acupuncture.

4.2 Subjective assessment A quality of life questionnaire (FACT/GOG-NTX v4) will be filled in by patients at enrolment, commencement, at the 6th session and at the end of 10 sessions of acupuncture.

4.3 Scoring With both objective and subjective assessment, a Total Neuropathy Score can be calculated at each time point as a quantitative measurement of the severity of PN

5. Statistical considerations The statistical analysis specifies that a lower limit of the two-sided 90 percent confidence interval for the overall positive response that exceeded 10 percent would be considered to be evidence of significant efficacy of acupuncture in retarding Bortezomib or thalidomide induced PN. Allowing a confidence interval width of 30%, the sample size needed will be 34 patients. To allow for a 10% drop-out, we plan to recruit a total of 40 patients

ELIGIBILITY:
Inclusion Criteria:

1. Age > 21 years and have a diagnosis of a plasma cell dyscrasia or lymphoma.
2. Patients must have neuropathy greater or equal to 2 according to CTCAE v 3.0 scale in spite of adequate duration (at least 3 weeks) of previous treatment with Gabapentin or Pregabalin or are unable to tolerate these drugs. Patients receiving any of these drugs must remain on the same medications throughout the study period; however, minor adjustments in dosage are allowed.

3. The patient's current or previous treatment must include bortezomib or thalidomide

4. ECOG Performance Status of 0, 1, or 2

Exclusion Criteria:

1. Local infection at or near the acupuncture site. (Although acupuncture is a minimally invasive procedure, patients will be excluded if there is an indication of active infection.)
2. Thrombocytopenia (platelet counts < 50x 109/L) on the day of acupuncture session
3. Deformities that could interfere with accurate acupuncture point location or out of energy pathway as defined by traditional acupuncture theory.
4. Concurrent use of anticoagulation agents.
5. Known coagulopathy and taking heparin (including low molecular weight heparin) or warfarin at any dose. Patients on aspirin or non-steroidal anti-inflammatories are allowed to participate.
6. Persistent absolute neutrophil counts of < 1 x 109/L
7. Active CNS disease.
8. Patients having a cardiac pacemaker.
9. Currently pregnant or lactating females.
10. Severe diabetic neuropathy or neuropathy related to HIV.
11. Previous acupuncture treatment for any indication within 30 days of enrollment.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2012-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Improvement in peripheral neuropathy | within the 5 weeks of acupuncture treatment

CONTACTS AND LOCATIONS:
Overall Officials: Yeh-Ching Linn, MBBS, MRCP, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore